CLINICAL TRIAL: NCT05713942
Title: Concussion Assessments in Football Competitions Participating in the IFAB's Permanent Concussion Substitution Trial
Brief Title: Concussion Assessments in Football
Status: Enrolling by invitation | Type: Observational
Sponsor: Federation Internationale de Football Association (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 006
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Concussion; Brain Concussion; Post-Concussion Symptoms; TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Sport Concussion Assessment Tool 5th Edition (SCAT5) — The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals 13 years old or older, who are suspected of having sustained a sports-related concussion. It comprises a neuropsychological test battery that assesses attention and memory function through 8 different domains 1) Symptom number, 2) Symptom severity, 3) Orientation, 4) Immediate memory, 5) Concentration, 6) Neurological examination, 7) Balance errors, 8) Delayed recall.
Diagnostic Test: The Immediate Post-Concussion Assessment and Cognitive Testing tool version 4 (ImPACT) — The ImPACT is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussion in individuals ages 12-80 years

SUMMARY:
Diagnosing and determining the severity of a sports-related concussion immediately on- or off-field is challenging, especially because clinical signs can evolve minutes to hours after the mechanism of injury. Hence, repeated follow-up and serial assessments of a player are recommended following such an injury.

Current advice, when a player sustains a confirmed or suspected concussive injury, is to remove them from play immediately and not return to competition or unrestricted training until signs and symptoms have been managed as per relevant guidelines. To support this decision the International football Association Board has introduced a trial allowing an additional permanent concussion substitution in participating competitions. Follow-up assessment of concussion incidents is recommended to include the Sport Concussion Assessment Tool 5th Edition. For further assessment of neurocognitive deficits and to inform return to play decisions, it is recommended that a computerised assessment is also adopted, such as the Immediate Post-Concussion Assessment and Cognitive Testing tool.

The aims of this study are:

1. To determine the incidence of head trauma and use of concussion substitutions in football competitions that are participating in the IFAB's permanent concussion substitution trial.
2. To evaluate the immediate severity of reported concussion signs and symptoms for football players with a confirmed or suspected concussion.
3. To evaluate the ability of neurocognitive assessments completed post-incident to inform the clinical diagnosis of concussion.

DETAILED DESCRIPTION:
1 INTRODUCTION

Concussions represent a subset of traumatic brain injury (TBI), pragmatically described as a "traumatically induced transient disturbance of brain function caused by a complex physiological process". A sports-related concussion (SRC) can result in substantially different outcomes, ranging from no detectable effects to transient functional impairments or even life-threatening complications. While the immediate effects of most concussions are short-lived, typically resolving within days, athletes who continue to play following a concussive event may increase their risk of developing short-, medium-, and long-term consequences.

TBI and SRC in football have received increased attention from medical and scientific communities, sports organisations, legislators, the media, as well as the general population. Consistency in the identification of concussed footballers and their subsequent management and rehabilitation has received particular focus. It is apparent that the management of suspected and confirmed concussive events are prominent and contentious issues in football. Incidence of SRC varies considerably across studies, which may be largely due to methodological differences. During 51 FIFA affiliated tournaments and 4 Olympic Games from 1998 to 2012, 3944 injuries were reported by the Team Physicians, of which 577 (15%) affected the head or neck. Eighty-one injuries (2% of all injuries) were given the diagnosis of concussion. It is pertinent to more accurately establish the incidence of head trauma and concussive injuries as allows risk exposure to be better understood.

Diagnosing and determining the severity of a SRC immediately on- or off-field is challenging, especially because clinical signs can evolve minutes to hours after the mechanism of injury. Hence, repeated follow-up and serial assessments of a player are recommended following such an injury. Combined injuries of the central and peripheral nervous systems are frequent, determining the locus of injury and therefore underlying explanation for symptoms is difficult and often not possible on- or off-field requiring a more focussed examination. Thus, the diagnosis and estimation of injury severity on- or off-field is a major challenge for the personnel performing an assessment. Specific predictors of injury severity, prognosis and the likely temporal resolution of symptoms are yet to be determined in a football population. Nevertheless, an immediate, targeted and standardised assessment approach to support clinical decision-making is of great importance, and despite unanswered research questions in this specific population, it does help to guide the management approach.

Current advice, when a player sustains a confirmed or suspected concussive injury, is to remove them from play immediately and not return to competition or unrestricted training until signs and symptoms have been managed as per relevant guidelines. To support this decision the International football Association Board has introduced a trial allowing an additional permanent concussion substitution in participating competitions. Follow-up assessment of concussion incidents is recommended to include the Sport Concussion Assessment Tool 5th Edition (SCAT5). The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals aged 13 years or older, who are suspected of having sustained an SRC. It comprises a neuropsychological test battery that assesses attention, memory and neurological function through 8 different domains. It's particular utility is in the immediate assessment of the athlete and in the first 3-5 days following the incident, subsequently it can be used to track symptom resolution. For further assessment of neurocognitive deficits and to inform return to play decisions, it is recommended that a computerised assessment is also adopted. The Immediate Post-Concussion Assessment and Cognitive Testing tool version 4 (ImPACT) is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussed individuals aged 12-80 years. The application of these two assessment modalities and their ability to inform clinical-decision making regarding concussion diagnosis in a football population has not been considered before, this includes whether their utility differs if compared to individual or normative baseline neurocognitive assessment values.

2 PROJECT OBJECTIVES AND DESIGN 2.1 Hypothesis and primary objective

1. The primary aim is to determine the incidence of head trauma and use of concussion substitutions in football competitions that are participating in the IFAB's permanent concussion substitution trial.
2. To evaluate the immediate severity of reported concussion signs and symptoms for football players with a confirmed or suspected concussion.
3. To evaluate the ability of neurocognitive assessments completed post-incident to inform the clinical diagnosis of concussion.

Our hypothesis is that there will be a variation in concussion severity with most incidents resulting in minor symptoms only, but still to a level where these can be detected in the post-incident assessments compared to baseline values and therefore inform the clinical diagnosis made.

2.2 Primary and secondary endpoints

1. To compare the concussion symptoms and domain scores post-incident with individual player baseline values, if available, otherwise normative values will be used.
2. To determine the temporal relationship of concussion signs and symptoms following the injury incident until full return to play.
3. If players consent, to assess mechanisms of concussion injury through video analysis of the incidents and compare these features to post-incident assessments.

2.3 Project design

International multi-centre prospective cohort study.

3 PROJECT POPULATION AND STUDY PROCEDURES 3.1 Study background

The International Football Association Board (IFAB) have initiated a trial of implementing additional permanent concussion substitutions (APCS) for actual or suspected concussions as of January 2021. This has been facilitated by making amendments to Law 3 in the rules of the game. With this Law there are 2 protocols (Appendix 1), with National Football Associations able to adopt one in a competition. The protocols are:

* Protocol A: enables one "concussion substitute" per team and no additional substitute for the opposing team
* Protocol B: enables two "concussion substitutes" per team and an additional substitute for the opposing team

All 211 FIFA member associations (National Football Associations) are invited to participate in this trial. Participation is voluntary. The National Football Associations can participate with as many competitions as they wish and adopt one of the above protocols per competition. Competitions refer to different levels of organized leagues, as well as cup tournaments. Additionally, competitions organized by FIFA, such as the FIFA World Cup, are automatically participating in the trial.

In agreeing to be a part of the trial, the National Football Associations must also supply FIFA with feedback information so that the Law change can be accurately reviewed. This feedback is divided into 3 categories and includes competition information, in-game information, and medical information. The medical information requirements are outlined in the Concussion Substitutes Trial Medical Assessment and include baseline neurocognitive assessments (SCAT5 and ImPACT).

3.2 Project population, inclusion and exclusion criteria

All National Football Associations participating in the IFAB's additional permanent substitutions trial are requested to provide post incident medical assessment data from appropriately consented players (explained below) within their competitions according to the following eligibility criteria

Inclusion criteria Male and female football players from teams in a competition participating in the concussion substitution trial.

Player assessed by medical personnel proficient in the assessment of concussion symptoms (medical doctor, physiotherapist, or other healthcare professional appropriately certified).

Exclusion criteria Players less than 18 years of age. Players with a current suspected or confirmed concussion Any other sustained injury that requires hospital admission

3.2 Recruitment, screening, and informed consent procedure

The IFAB additional permanent substitutions trial is expected to run from January 2021 to August 2023 with potential for extension. All teams from participating competitions will be contacted and invited to participate. Contact information is gathered from the respective competition organisers.

All players who experience a concussion incident during the trial period will receive oral and written information about the research project. The study information will be translated and be available in the four official FIFA languages; English, German, Spanish, and French. Additional translations will be discussed on an individual basis with the respective National Football Association. The players will have the opportunity to provide consent in two parts:

1. Consent to participate with standard concussion medical assessment data, which is coded to ensure complete anonymisation
2. Consent to participate with video footage analysis of the concussion incident (which allows identification of the player), combining this information with post-injury concussion medical assessments

Players do not have to consent to both parts of the research project. A written informed consent form will be gathered for each part of the project.

3.3 Study procedures

The study is a prospective cohort study, it will run for the same period as the IFAB additional permanent substitutions trial. All concussion substitutions occurring during the trial period are registered online through the FIFA data platform by the respective Team or National Football Association. The research project is considered to have minimal risk, risk category A according to art. 7 (HRO). No procedures are required from participants as a direct result of the research project as they will follow standard guidelines on assessment according to their individual setting. Participants are therefore not exposed to any additional health risks from participation in the research and there is only a minimal burden in registration of assessments.

Players who have experienced a suspected or confirmed concussive injury during a competitive match will be asked to participate in the research project. There is currently no diagnostic test or biomarker that determines a diagnosis of SRC2, the presence or absence of this diagnosis is therefore determined by the medical professional with primary responsibility of the player's care. Medical professionals are requested to complete the Concussion Substitute Trials Medical Assessment. Additionally, follow-up concussion assessments using the SCAT5 and/or ImPACT performed by a healthcare professional proficient in the assessment of concussion symptoms should be performed at specific timepoints following the injury. These assessments should be uploaded on to the FIFA data platform with the associated baseline neurocognitive assessments (SCAT5 and ImPACT) if these have been completed.

SCAT5 The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals 13 years old or older, who are suspected of having sustained a sports-related concussion. It comprises a neuropsychological test battery that assesses attention and memory function through 8 different domains 1) Symptom number, 2) Symptom severity, 3) Orientation, 4) Immediate memory, 5) Concentration, 6) Neurological examination, 7) Balance errors, 8) Delayed recall.

The time required for assessment using the SCAT5 is minimum 10 min. The only equipment required for the tester is a watch or timer.

Reliability Reliability of the SCAT5 has been tested in other settings. In 62 professional ice hockey players the two-week test-retest reliability of the SCAT5 baseline scores varied from poor to high. There was considerable individual variability and most players have notable short-term fluctuation on performance even if uninjured. The study calculated stability coefficients using Spearman's r for the separate SCAT5 domains; Symptom number r=0.85, p<0.001, Symptom severity r=0.84, p<0.001, Orientation (0-30) r=-0.14, p = 0.283, Immediate memory r=0.40, p=0.001, Concentration r=0.62, p<0.001, Delayed recall (0-10) r=0.45, p<0.001, Balance errors r=0.40, p=0.001.

The SCAT5 document is submitted separately.

ImPACT The ImPACT is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussion in individuals ages 12-80 years.

The ImPACT test should be performed in an environment which must be quiet and distraction-free, with no phones or other devices available. The test person should sit comfortably at a table or desk with a flat, hard surface. A computer with a keyboard and a mouse or a trackpad is used for the test with all other programs and browsers tabs closed. The ImPACT provides 5 composite scores for verbal memory, visual memory, visual motor-speed, reaction time, and impulse control, as well as a total symptom score. Two-factor scores for memory and speed are also provided.

The time required to perform the ImPACT assessment is maximum 45 min. The equipment needed is a computer with keyboard, and mouse/trackpad, and access to the online tool (provided free for all participants through FIFA).

Reliability A meta-analysis of the reliability of the ImPACT has shown moderate to substantial test-retest reliability of the IMPACT domains with pooled intraclass correlation coefficients (ICCs): verbal memory: 0.52 (95%CI 0.44-0.66), visual memory: 0.56 (95%CI 0.48-0.62), visual-motor speed: 0.7 (95%CI 0.72-.0.81), and reaction time: 0.65 (95%CI 0.59-0.71).16 No differences were identified based on average length of the test-retest interval or between athletes and the general population.

Further information on the ImPACT can be found on https://impacttest.com/ and https://impactconcussion.com/.

Video analysis Given that incident video footage will enable players to be able identified, all players will need to provide additional informed consent, prior to uploading this identifiable information regarding. If there is video footage of the incident available, this can be uploaded directly on to the data platform. Alternatively, broadcast footage will be sought for analysis.

A standardized video analysis protocol will be adopted to facilitate consistent reporting of injury mechanism and related match-specific features. This will incorporate the international consensus definitions of video signs of concussion.

3.4 Withdrawal and discontinuation

Individual participants can withdraw their data from this study without giving a reason at any time prior to analysis completion.

Participating competitions can withdraw from the IFAB APCS trial at any time without giving a reason. In such circumstance, the IFAB must be notified in writing. In case the competition organisers commit a breach of the signed declaration, the IFAB can withdraw the permission to participate in the trial. In case of any withdrawal from the trial the collected data prior to withdrawal will be kept, except if requested otherwise.

4 STATISTICS AND METHODOLOGY 4.1. Statistical analysis plan Concussion assessments Concussion assessment results will be summarized using descriptive statistics (mean, standard deviation, median, interquartile range) according to their distribution at the specified timepoints when they were completed following the injury. The rate of compliance with the aspects of the assessments will be reported.

Post-concussion incident assessment values are compared to individual baseline assessments when available and to normative reference values in football players. Baseline data obtained in this study will be combined with baseline data obtained as part of a connected study within the same project (BASEC application number 2022-00016), it will be the results of this study which inform the normative reference values in football players. Comparisons to baseline assessments will be made for each assessment domain and at each specified post-incident assessment timepoint. The baseline data will also be used to create cut-off scores, to assist the diagnostic decision-making process. The appropriateness of adopting the 10th percentile as a cut-off in line with previous research conducted in professional ice hockey, will be considered.

The data will be assessed for normality and appropriate data transformations or non-parametric tests will be used if necessary. Depending on distribution dependent-tests and independent t-tests or Mann-Whitney U test and Wilcoxon Signed Ranks tests will be used for the group comparisons. Cohen's d will be used to estimate effect sizes, with effects sizes interpreted as small (d = 0.2), moderate (d = 0.5), and large (d = 0.8).19 The level of statistical significance will be set at p-value of <0.05. Receiver operating characteristic (ROC) curves will be calculated to examine the classification accuracy for concussed and non-concussed players. In addition, dichotomous data (e.g., diagnosis of concussion) will be analysed using log-binomial regression models. Adjusting for baseline SCAT5 and ImPACT scores, these models will be used to calculate relative risks and 95% confidence intervals.

Time to event data, including resolution of recorded symptoms and return to play duration will be analysed using the log-rank test with a Cox Proportional Hazard model used to calculate hazard ratios, if the assumptions of proportionality are met.

Sample size Due to the nature of the pathology being investigated, sample size is difficult to predict or guarantee. The aim is to include all available data during the trial period with a target of 100 players with concussion incidents, which is considered feasible based on the international multi-centre nature and length of trial period. Based on reported values from professional ice hockey it can be expected that the smallest differences on the SCAT5 components will be for immediate memory, concentration, and delayed recall. Informed by this research, a difference in the concentration score of 0.4 between baseline and post-incident assessment may be expected. With a baseline mean of 3.5, an average standard deviation of 0.9, an alpha value of 0.05, and a power of 0.8, 81 concussion incidents assessments would be required for analysis.

Video analysis All concussions with video footage and player consent will be included. A standardised protocol will be adopted to analyse all footage received. Simple descriptive statistics will be applied to provide an overview of frequencies of the different concussion injury mechanisms. Video analysis variables will be compared to concussion assessment findings (e.g. severity of symptoms) and time to event data (e.g. resolution of symptoms, return to play duration), if possible, to understand if any correlation exists.

4.2. Handling of missing data Every attempt will be made to ensure a complete dataset, with Medical Staff being contacted if submissions are not complete. Potential missing data will be excluded from analysis and reported accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Male and female football players from teams in a competition participating in the concussion substitution trial.
* Players with a current suspected or confirmed concussion.
* Player assessed by medical personnel proficient in the assessment of concussion symptoms (medical doctor, physiotherapist, or other healthcare professional appropriately certified).

Exclusion Criteria:

- Players less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any football player playing an official match in a competition participating in the IFAB's permanent concussion substitution trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concussion incident | January 1st 2021 to August 31st 2023
  Any incident of a suspected or actual concussion occurring in a football match where the permanent concussion substitution was or could have been used.

SECONDARY OUTCOMES:
SCAT5 assessment | Baseline (noninjured), and immediate, +1 day, and +3 days post-concussion incident
  The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals 13 years old or older, who are suspected of having sustained a sports-related concussion. It comprises a neuropsychological test battery that assesses attention and memory function through 8 different domains 1) Symptom number, 2) Symptom severity, 3) Orientation, 4) Immediate memory, 5) Concentration, 6) Neurological examination, 7) Balance errors, 8) Delayed recall
IMPACT assessment | Baseline (noninjured), and immediate, +3 days, and +6 days post-concussion incident
  The ImPACT is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussion in individuals ages 12-80 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Serner, PhD, Principal Investigator — Fédération Internationale de Football Association
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No